CLINICAL TRIAL: NCT04174235
Title: Fetal Congenital Anomalies Among Egyptian Pregnant Women Attending University Hospital
Brief Title: Prevalence of Fetal Congenital Anomalies Among Pregnant Women Attending University Hospital
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Associate Professor in Obstetrics and Gynecology Department, Beni-Suef University
Other Study IDs: Beni-Suef 18
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Fetal Anomaly
Keywords: Fetal anomalies
MeSH Terms: conditions — Congenital Abnormalities | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound scan — A full history taking was obtained according European surveillance of congenital anomalies EURO-CAT core data. All women underwent abdominal and transvaginal US (Toshiba Xario 200 unit)

SUMMARY:
Congenital anomalies occur in 2-3% of births. They account for 20-30% of perinatal deaths. The aim is to assess the prevalence of fetal malformations in pregnant women attending University hospital

DETAILED DESCRIPTION:
This prospective cohort study of 20225 pregnant women attended Obstetrics Department of Beni-Suef University Hospital during period (January 2016 to January 2019). A full history taking was obtained according European surveillance of congenital anomalies EURO-CAT core data. All women underwent abdominal and transvaginal US (Toshiba Xario 200 unit): ▪ Females presented early in first trimester were scheduled for routine first trimester scan in accordance with international society of ultrasound in obstetrics and gynecology guidelines. ▪ Females presented early in second trimester were scheduled for a routine second trimester scan. ▪ Females presented afterwards, had a routine ultrasound scan for fetal malformations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy

Exclusion Criteria:

* Medical conditions, chronic drug intake.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women attended Obstetrics and Gynecology Department of Beni-Suef University Hospital during the period (January 2016 to January 2019)
Sampling Method: Non-Probability Sample
Enrollment: 20225 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
prevalence of fetal malformations in pregnant women | Up to 37 weeks
  Females presented early in first trimester were scheduled for routine first trimester scan in accordance with international society of ultrasound in obstetrics and gynecology guidelines. ▪ Females presented early in second trimester were scheduled for a routine second trimester scan. ▪ Females presented afterwards, had a routine ultrasound scan for fetal malformations.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busby A, Abramsky L, Dolk H, Armstrong B; Eurocat Folic Acid Working Group. Preventing neural tube defects in Europe: population based study. BMJ. 2005 Mar 12;330(7491):574-5. doi: 10.1136/bmj.330.7491.574. No abstract available. PMID 15760997
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442